CLINICAL TRIAL: NCT05578456
Title: Effect of Prednisone and Aspirin on Pregnancy Outcomes After Embryo Transfer Among Patients With Thyroid Autoimmunity: a Randomized Clinical Trial
Brief Title: Effect of Prednisone and Aspirin on IVF-ET Outcome Among Patients With Thyroid Autoimmunity
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Women & Children's Hospital (Other); Jinhua People's Hospital (Other); Jiaxing Maternity and Child Health Care Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0513
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Thyroiditis, Autoimmune; Infertility
MeSH Terms: conditions — Thyroiditis, Autoimmune; Infertility | interventions — Prednisone; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisone and aspirin (Experimental)
  Interventions: Drug: Prednisone and Aspirin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone and Aspirin — prednisone 10 mg and aspirin 75-100mg per day per os
  Arms: prednisone and aspirin
Drug: Placebo — placebo 2 starch tablets per day per os
  Arms: placebo

SUMMARY:
This trial was a 1:1 (active:placebo) randomized, double-blind, placebo-controlled trial to evaluate the safety and efficacy of prednisone and aspirin for the in vitro fertilization and embryo transfer outcome among patients with thyroid autoimmunity.

ELIGIBILITY:
Inclusion Criteria:

1. TPOAb>34IU/ml and/or TgAb>115IU/ml
2. ≥5 follicles with average diameter lager than 14 mm at trigger day
3. ≥5 oocytes retrieved
4. for frozen embryo transfer, at least 2 cleavage stage embryos, among which at least one morphologically good quality embryo, or at least 1 morphologically good quality embryo in blastocyst stage
5. age: 20-38 years old
6. Patients whose written ICF approved by the EC has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.

meet item 1, 5, 6, and one of item 2, 3, 4.

Exclusion Criteria:

* hyperthyroidism
* intrauterine adhesion
* with endometrium thickness less than 6mm
* uterine malformation
* PGT
* with other autoimmune diseases need glucocorticoid or aspirin treatment
* gluacoma
* gastric ulcer

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 540 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 3-5 weeks after embryo transfer
  ultrasound visualization of the gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Min Jin, Doctor, Principal Investigator — Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided